CLINICAL TRIAL: NCT06262815
Title: The Utility of Treatment With Nasogastric Tube Placement for Small Bowel Obstruction in Adult Patients in the Emergency Department; an Observational Multicenter Study
Brief Title: The Utility of Treatment With Nasogastric Tube Placement for Small Bowel Obstruction
Acronym: NGTUBE-OBS
Status: Recruiting | Type: Observational
Sponsor: Daniel Wilhelms (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Daniel Wilhelms, Head of Research, Department of Emergency Medicine, Associate Professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Other Study IDs: 2023-06806-01
Record Dates: First submitted 2023-12-29; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Small Bowel Obstruction; Frailty; Nasogastric Tube
Keywords: Small bowel obstruction; nasogastric tube; pain; mortality; morbidity; frailty
MeSH Terms: conditions — Frailty; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with nasogastric tube treatment: Adult patients with diagnosed small bowel obstruction in the Emergency Department for a nasogastric tube was placed
  Interventions: Procedure: Nasogastric tube placement
- Patients without nasogastric tube treatment: Adult patients with diagnosed small bowel obstruction in the Emergency Department for no nasogastric tube was placed
  Interventions: Procedure: Nasogastric tube placement
- Patients living with frailty: Subgroup of patients, with small bowel obstruction in the Emergency Department over 65 years of age with a clinical frailty score of >4.
  Interventions: Diagnostic Test: Clinical Frailty Scale
- Patients not living with frailty: Subgroup of patients, with small bowel obstruction in the Emergency Department over 65 years of age with a clinical frailty score of <5.
  Interventions: Diagnostic Test: Clinical Frailty Scale

INTERVENTIONS:
Procedure: Nasogastric tube placement — Conventional nasogastric tube placement done for decompression of small bowel obstruction
  Groups: Patients with nasogastric tube treatment; Patients without nasogastric tube treatment
Diagnostic Test: Clinical Frailty Scale — The scale described by Rockwood et al. categorizing patients >65 years of age on a 9 item scale depending on the frailty.
  Groups: Patients living with frailty; Patients not living with frailty

SUMMARY:
Small bowel obstruction (SBO) occurs when the normal movements of the small bowel is obstructed, most commonly due to adhesion related to previous abdominal surgery. This may cause strangulation of the small bowel with reduced blood flow which is a surgical emergency requiring prompt treatment in the operating room. If there are no signs of strangulation or ischemia of the bowel at the time of diagnosis, international guidelines recommend initial treatment with intravenous fluids and nasogastric tube placement. However, there is emerging debate regarding non-selective treatment with nasogastric tube placement in patients with SBO. This management started around 1930 as a means to reduce pain in patients with SBO, in conjunction with other additions to management, like intravenous fluids. However the effect and utility of routine nasogastric tube placement have not been prospectively evaluated. There are a total of three retrospective observational studies in the past decade with a total of 759 patients where 292 (36%) were managed without a nasogastric tube. There was no difference in the rates of conservative treatment failure (requiring surgery), complications (vomiting, pneumonia) or mortality between patients receiving a nasogastric tube and those who didn't. However, the retrospective design of these studies limits their validity. Furthermore, nasogastric tube placement has been shown to be one of the more painful interventions patients may experience in-hospital. This calls into question the patient benefit of routine nasogastric tube placement in patients with SBO and further studies are needed to discern the utility of this intervention.

Definitive treatment for SBO is surgical adhesiolysis but there is debate regarding the timing of surgery, particularly in older adults. A large proportion of patients may be managed conservatively with oral contrast and repeated radiological evaluation and the obstruction will resolve in many patients within 24 to 48 hours. This timeframe is dependent on factors related to the disease itself as well as patient related factors like previous surgery and comorbidities. Older patients are at high risk for complications but current available data is insufficient to inform practice in this population. Frailty, a state of increased vulnerability and susceptibility to adverse events, has been shown to be an independent prognosticator in older adults in the Emergency Department(ED) and suggested as a potential measure to risk stratify older adults with SBO. However to the authors knowledge there is no available data on frailty in older adults with SBO and only one prospective observational trial looking at older adults with SBO. Despite SBO being one of the most common surgical emergencies in older adults.

To investigate the potential benefit of nasogastric tube placement in patients with SBO and the ability of frailty to prognosticate outcomes in older adults better evidence is needed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed small bowel obstruction
* Age 18 or older

Exclusion Criteria:

* Abdominal surgery within 7 days
* Not able to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting any of the following Emergency Departments in Sweden:
  * Linköping University Hospital
  * Motala Lasarett
  * Vrinnevisjukhuset Norrköping
  * Sundvalls Lasarett
  * Skåne University Hospital Malmö
  * Skåne University Hospital Lund
  * Sahlgrenska University Hospital Sahlgrenska
  * Sahlgrenska University Hospital Östra
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain at Emergency Department discharge | at Emergency Department Discharge, assessed up to 48 hours
  self-reported Pain on a Numeric Rating Scale from 0 to 10 were higher is worse

SECONDARY OUTCOMES:
Nausea at Emergency Department discharge | at Emergency Department discharge, assessed up to 48 hours
  Nausea as self-reported by patients on a numeric rating scale from 0 to 10 were higher is worse
Hospital Length of Stay | Up to 90 days from inclusion
  Duration of days spent in the hospital by patients with Small Bowel obstruction admitted from the Emergency Department
Mortality | up to 90 days from inclusion
  Mortality of any cause
Admission for Small bowel obstruction | up to 365 days from inclusion in the study
  Any admission to a hospital in Sweden with a primary discharge diagnosis of small bowel obstruction
Emergency Surgery | up to 30 days from inclusion
  Any emergency operation
Emergency Department Length of Stay | up to 7 days from inclusion
  Length of stay, defined as the time from registration in the Emergency Department to discharge from the Emergency Department at the visit of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Wilhelms, PhD, Principal Investigator — Linkoeping University
Locations (8):
- Sweden (8):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Östra sjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Skånes Universitetssjukhus, Malmo
  - Lasarett i Motala, Motala
  - Vrinnevisjukhuset, Norrköping
  - Sundsvalls sjukhus, Sundsvall
  - Akutmottagningen US Östergötland, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided
Limited (providing full anonymization) data may be provided to other researchers

REFERENCES:
- [Background] Elliott A, Taub N, Banerjee J, Aijaz F, Jones W, Teece L, van Oppen J, Conroy S. Does the Clinical Frailty Scale at Triage Predict Outcomes From Emergency Care for Older People? Ann Emerg Med. 2021 Jun;77(6):620-627. doi: 10.1016/j.annemergmed.2020.09.006. Epub 2020 Dec 13. PMID 33328147
- [Background] Rueegg M, Nissen SK, Brabrand M, Kaeppeli T, Dreher T, Carpenter CR, Bingisser R, Nickel CH. The clinical frailty scale predicts 1-year mortality in emergency department patients aged 65 years and older. Acad Emerg Med. 2022 May;29(5):572-580. doi: 10.1111/acem.14460. Epub 2022 Apr 23. PMID 35138670
- [Background] Kaeppeli T, Rueegg M, Dreher-Hummel T, Brabrand M, Kabell-Nissen S, Carpenter CR, Bingisser R, Nickel CH. Validation of the Clinical Frailty Scale for Prediction of Thirty-Day Mortality in the Emergency Department. Ann Emerg Med. 2020 Sep;76(3):291-300. doi: 10.1016/j.annemergmed.2020.03.028. Epub 2020 Apr 24. PMID 32336486
- [Background] Ozturk E, van Iersel M, Stommel MM, Schoon Y, Ten Broek RR, van Goor H. Small bowel obstruction in the elderly: a plea for comprehensive acute geriatric care. World J Emerg Surg. 2018 Oct 20;13:48. doi: 10.1186/s13017-018-0208-z. eCollection 2018. PMID 30377439
- [Background] Koh A, Adiamah A, Chowdhury A, Mohiuddin MK, Bharathan B. Therapeutic Role of Water-Soluble Contrast Media in Adhesive Small Bowel Obstruction: a Systematic Review and Meta-Analysis. J Gastrointest Surg. 2020 Feb;24(2):473-483. doi: 10.1007/s11605-019-04341-7. Epub 2019 Aug 13. PMID 31485900
- [Background] Springer JE, Bailey JG, Davis PJ, Johnson PM. Management and outcomes of small bowel obstruction in older adult patients: a prospective cohort study. Can J Surg. 2014 Dec;57(6):379-84. doi: 10.1503/cjs.029513. PMID 25421079
- [Background] Hajibandeh S, Hajibandeh S, Panda N, Khan RMA, Bandyopadhyay SK, Dalmia S, Malik S, Huq Z, Mansour M. Operative versus non-operative management of adhesive small bowel obstruction: A systematic review and meta-analysis. Int J Surg. 2017 Sep;45:58-66. doi: 10.1016/j.ijsu.2017.07.073. Epub 2017 Jul 17. PMID 28728984
- [Background] Peacock O, Bassett MG, Kuryba A, Walker K, Davies E, Anderson I, Vohra RS; National Emergency Laparotomy Audit (NELA) Project Team. Thirty-day mortality in patients undergoing laparotomy for small bowel obstruction. Br J Surg. 2018 Jul;105(8):1006-1013. doi: 10.1002/bjs.10812. Epub 2018 Mar 30. PMID 29603126
- [Background] Kuo YW, Yen M, Fetzer S, Lee JD. Reducing the pain of nasogastric tube intubation with nebulized and atomized lidocaine: a systematic review and meta-analysis. J Pain Symptom Manage. 2010 Oct;40(4):613-20. doi: 10.1016/j.jpainsymman.2010.01.025. Epub 2010 Aug 3. PMID 20678892
- [Background] Morrison RS, Ahronheim JC, Morrison GR, Darling E, Baskin SA, Morris J, Choi C, Meier DE. Pain and discomfort associated with common hospital procedures and experiences. J Pain Symptom Manage. 1998 Feb;15(2):91-101. PMID 9494307
- [Background] Berman DJ, Ijaz H, Alkhunaizi M, Kulie PE, Vaziri K, Richards LM, Meltzer AC. Nasogastric decompression not associated with a reduction in surgery or bowel ischemia for acute small bowel obstruction. Am J Emerg Med. 2017 Dec;35(12):1919-1921. doi: 10.1016/j.ajem.2017.08.029. Epub 2017 Aug 15. PMID 28912083
- [Background] Edlich RF, Woods JA. Wangensteen's transformation of the treatment of intestinal obstruction from empiric craft to scientific discipline. J Emerg Med. 1997 Mar-Apr;15(2):235-41. doi: 10.1016/s0736-4679(96)00351-4. PMID 9144067
- [Background] Klingbeil KD, Wu JX, Osuna-Garcia A, Livingston EH. Management of small bowel obstruction and systematic review of treatment without nasogastric tube decompression. Surg Open Sci. 2022 Nov 7;12:62-67. doi: 10.1016/j.sopen.2022.10.002. eCollection 2023 Mar. PMID 36992798
- [Background] Shinohara K, Asaba Y, Ishida T, Maeta T, Suzuki M, Mizukami Y. Nonoperative management without nasogastric tube decompression for adhesive small bowel obstruction. Am J Surg. 2022 Jun;223(6):1179-1182. doi: 10.1016/j.amjsurg.2021.11.029. Epub 2021 Dec 2. PMID 34872712
- [Background] Ten Broek RPG, Krielen P, Di Saverio S, Coccolini F, Biffl WL, Ansaloni L, Velmahos GC, Sartelli M, Fraga GP, Kelly MD, Moore FA, Peitzman AB, Leppaniemi A, Moore EE, Jeekel J, Kluger Y, Sugrue M, Balogh ZJ, Bendinelli C, Civil I, Coimbra R, De Moya M, Ferrada P, Inaba K, Ivatury R, Latifi R, Kashuk JL, Kirkpatrick AW, Maier R, Rizoli S, Sakakushev B, Scalea T, Soreide K, Weber D, Wani I, Abu-Zidan FM, De'Angelis N, Piscioneri F, Galante JM, Catena F, van Goor H. Bologna guidelines for diagnosis and management of adhesive small bowel obstruction (ASBO): 2017 update of the evidence-based guidelines from the world society of emergency surgery ASBO working group. World J Emerg Surg. 2018 Jun 19;13:24. doi: 10.1186/s13017-018-0185-2. eCollection 2018. PMID 29946347
- [Background] Long B, Robertson J, Koyfman A. Emergency Medicine Evaluation and Management of Small Bowel Obstruction: Evidence-Based Recommendations. J Emerg Med. 2019 Feb;56(2):166-176. doi: 10.1016/j.jemermed.2018.10.024. Epub 2018 Dec 6. PMID 30527563